CLINICAL TRIAL: NCT00148655
Title: A Randomized Trial for Educational Interventions for Patients With DCIS Actually Making Treatment Decisions
Brief Title: Educational Interventions for Patients With DCIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Eric Winer, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 02-331
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: DCIS
Keywords: educational intervention; decision board; DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

INTERVENTIONS:
Device: Decision Board — Decision board that explains the risks and benefits of treatment options

SUMMARY:
The purpose of this study is to determine whether adding an educational intervention, in the form of a decision board, which outlines the risks and benefits of treatment options for DCIS, at the time of the first surgical consultation will improve decision making for women with DCIS.

DETAILED DESCRIPTION:
* The decision board explains the risks and benefits of mastectomy, excision and radiation, excision, radiation, and tamoxifen, excision alone, and excision without radiation and tamoxifen for women with DCIS.
* Patients will receive a decision board to take home for review. Two fifteen-minute telephone interviews will be conducted, one approximately one week after enrollment and one 2 months after enrollment.
* In the phone interviews, patients will asked to complete a brief survey. This survey will ask abou DCIS in general, the patient's treatment decisions, their feelings, as well as their experience with the decision board.
* This study will take about 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include women over the age of 25 with newly-diagnosed DCIS who are candidates for breast conserving therapy.
* Pathologic confirmation of DCIS without evidence of invasive breast cancer and mammograms showing a single suspicious focus without mammographic or clinical evidence of multicentricity.
* Patients that have not made a decision regarding management of DCIS
* Eligible for radiotherapy to breast
* Oral and written knowledge of English

Exclusion Criteria:

* Patients that have undergone mastectomy
* History of prior radiotherapy to the breast, scleroderma or systemic lupus erythematosus
* Clinically palpable disease in the axilla or contralateral breast cancer
* Co-morbidities that would render them ineligible for general anesthesia

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine the impact of an educational intervention on the decision-making in women with DCIS. | 3 years

SECONDARY OUTCOMES:
To assess the effect of an intervention on 1)satisfaction with decision-making, 2)knowledge of treatment options, 3)risk assessment, 4)treatment choice, 5)factors motivating treatment choice and 6)anxiety related to diagnosis. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts